CLINICAL TRIAL: NCT00267852
Title: An Observational Study To Evaluate The Clinical Remission In Early Aggressive Rheumatoid Arthritis (Artrite Reumatoide Precoce Aggressiva Italian Study)
Brief Title: Study Evaluating the Clinical Remission in Early Aggressive Rheumatoid Arthritis
Acronym: ARPA
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A-101749; B1801108
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Practice Guidelines as Topic; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1.0: As per routinary clinical practice
  Interventions: Other: as clinical practice

INTERVENTIONS:
Other: as clinical practice — Dosage, form, frequency and duration as per ordinary clinical practice
  Other Names: observational study

SUMMARY:
This is an observational prospective, multicenter study. The aim of the study is to evaluate how the Italian population of patients are treated with early aggressive RA, defined by the Italian Society of Rheumatology Guidelines, (GIARA Registry Study Group. Clin Exp Rheumatol 2003;21(Suppl. 31):S129-S132), in rheumatologic clinical practice and whether recent scientific evidence or new treatments available to rheumatologists can change their practice in a 2 year follow-up. The observation will primarily focus on the disease activity and clinical remission in patients who are receiving different treatment strategies. The primary goal is to define prevalence of clinical remission, according to the (Disease Activity Score) DAS 28 definition of clinical remission, in patients with early aggressive RA receiving different therapies at 1 year.

Secondary objective are assessment of:

* Prevalence of Remission at the second year
* Disease activity at the first and second year.
* ACR 20%, 50%, 70% response at the first and second year.
* Quality of Life in patients with or without remission at the first and second year
* Safety Evaluations

DETAILED DESCRIPTION:
It was expected that approximate 200 patients were enrolled in the study. Have been enrolled 152 patients. A Statistical Analysis Plan will contain a detailed description of criteria for valuable patients for analyses and a description of statistical analyses. In general, all patients who respond inclusion/exclusion criteria at baseline will be considered valuable for the study. The summaries will include descriptive statistics (mean, standard deviation, sample size) for the continuous parameters, and absolute frequencies and percentages for the remaining categorical parameters.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria Based On Clinical Practice of Aggressive RA

* Diagnosis of early aggressive RA in accordance with local guideline
* Disease duration < 2 years and at least six months since onset of symptoms
* Patients naïve to anti-TNFa drugs and DMARDs, including MTX, or assuming one or more DMARD without complete response

Exclusion Criteria:

Exclusion Criteria Based on Clinical Practice of Aggressive RA

* Patients should not be included in the study if they have participated in any interventional clinical trial within the previous 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early aggressive RA, who are treated in 15 specialized sites
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2006-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of clinical remission, according to the DAS 28 definition of clinical remission, in patients with early aggressive RA receiving different therapies at 1 year. | 12-24 months

SECONDARY OUTCOMES:
-Prevalence of Remission at the second year. | 12-24 months
Disease activity at the 1st and 2nd year | 12-24 months
ACR 20%, 50%, 70% response at the 1st and 2nd year | 12-24 months
QoL in patients with or without remission at the first and second year | 12-24 months
Safety Evaluations | 12-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- Italy (16):
  - Pfizer Investigational Site, Iesi, Ancona
  - Pfizer Investigational Site, Bari, Apulia
  - Pfizer Investigational Site, Napoli, Campania
  - Pfizer Investigational Site, Ferrara, Ferrara (FE)
  - Pfizer Investigational Site, Arenzano, GE
  - Pfizer Investigational Site, Rome, Lazio
  - Pfizer Investigational Site, Messina, Messina
  - Pfizer Investigational Site, Padua, Padova
  - Pfizer Investigational Site, Palermo, Palermo
  - Pfizer Investigational Site, Messina, Sicily
  - Pfizer Investigational Site, Siena, Siena
  - Pfizer Investigational Site, Pisa, Tuscany
  - Pfizer Investigational Site, Brescia
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Torino

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A-101749&StudyName=Study%20Evaluating%20the%20Clinical%20Remission%20in%20Early%20Aggressive%20Rheumatoid%20Arthritis